CLINICAL TRIAL: NCT05514496
Title: A First-in-Human, Open-Label, Dose Escalation and Expansion Study of Orally Administered NX-019 in Patients with Advanced, EGFR Mutant Cancer
Brief Title: A Study of NX-019 in Patients with Advanced, Epidermal Growth Factor Receptor (EGFR) Mutant Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nalo Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NT019-101
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: EGFR Mutation-Related Tumors
Keywords: NX-019; EGFR Mutant Cancer; CNS Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: NX-019 Dose Escalation (Experimental): Patients will be treated with NX-019 in multiple ascending cohorts.
  Interventions: Drug: NX-019
- Part 2: NX-019 Dose Expansion (Experimental): Patients will be treated with the REDs of NX-019 as determined in Part 1.
  Interventions: Drug: NX-019

INTERVENTIONS:
Drug: NX-019 — NX-019 will be administered orally.

SUMMARY:
This is a 2-part, first-in-human, open-label study to determine the safety and tolerability of NX-019 and preliminary efficacy in patients with locally advanced or metastatic epidermal growth factor receptor (EGFR)-mutant cancer.

DETAILED DESCRIPTION:
Part 1: The primary objective of Part 1 of this study is to evaluate the safety and tolerability of NX-019 and to determine the maximum tolerated dose (MTD)/Recommended Expansion Dose(s) (REDs).

Part 2: The primary objective of Part 2 of this study is to confirm the safety and tolerability of NX-019 at the REDs and, for each expansion cohort, the preliminary evidence of efficacy as measured by objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced, or metastatic EGFR-mutant cancer and has progressed on or are intolerant to all standard therapy.
* Patients with non-small cell lung cancer (NSCLC) harboring a mutation that is sensitive to osimertinib must have received osimertinib prior to enrollment.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (evaluable disease acceptable for dose escalation part of study).
* ≥18 years of age (or age of consent in in accordance with local law).
* Life expectancy ≥3 months.
* Adequate organ and bone marrow function.
* All patients will have a baseline magnetic resonance imaging (MRI) of the brain.
* Resolution of any clinically significant toxic effects of prior therapy to Grade 0 or 1 according to the National Cancer Institute CTCAE v5.0 (exception of alopecia and Grade 2 peripheral neuropathy).
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Willingness of men and women of reproductive potential to observe conventional and effective birth control methods with failure rates of <1% for the duration of treatment and for 6 months following the last dose of study treatment.
* A negative serum pregnancy test at Screening and a negative (serum or urine) pregnancy test within 72 hours before the first dose of study drug (female patients of childbearing potential only).
* Willing and able to give informed consent and comply with protocol requirements for the duration of the study.

Specific Inclusion Criteria for Expansion Cohorts:

To be eligible during the expansion part of the study, patients must meet the above inclusion criteria, and the criteria for 1 of the following cohorts:

Expansion Cohort 1:

* Patients with NSCLC with EGFR exon 19 deletions or exon 21 L858R mutations who have progressed on or after prior EGFR TKI therapy.

Expansion Cohort 2:

* Patients with NSCLC with EGFR ex20ins mutations, who are not suitable for, or are unwilling to receive available ex20ins mutation targeted therapy.

Expansion Cohort 3:

* Patients with NSCLC with EGFR mutations for which there is no current targeted therapy, (i.e., exclusion of exon 19, exon 21 L858R, and ex20ins mutation).

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in the study:

* Known C797X EGFR mutations or 1 or more known secondary drivers of disease.
* Disease requiring immediate palliative treatment with surgery or radiation therapy.
* Requirement for greater than 4 mg/day of dexamethasone (or equivalent) for management of CNS metastases.
* Received systemic anticancer chemotherapy, targeted agents, antibody therapy for cancer, immunotherapy for cancer, hormonal therapy or an investigational agent within 2 weeks or 5 half-lives (whichever is shorter) prior to start of study drug treatment.
* Major surgery within 3 weeks prior to start of study drug treatment.
* Radiation therapy within 4 weeks prior to start of study drug treatment.
* Severe or unstable cardiac conditions within 6 months prior to starting study drug treatment.
* Severe or unstable medical condition including uncontrolled diabetes or unstable psychiatric condition.
* Dependent on contact lenses (unable to wear eyeglasses) and unable to comply with ophthalmic guidance.
* History of interstitial lung disease, radiation pneumonitis which required systemic steroid therapy, or other significant lung disease.
* Another active malignancy within the previous 2 years except for localized cancers that are not related to the current cancer being treated, are considered cured, and, in the opinion of the Investigator, present a low risk of recurrence.
* Active infection requiring systemic therapy.
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) (i.e., hepatitis B surface antigen-positive), or hepatitis C virus (HCV) (i.e., detectable HCV ribonucleic acid [RNA]).
* Active gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or conditions that may impact drug absorption.
* Pregnant or breastfeeding.
* Is using a strong CYP3A inhibitor or inducer, and cannot refrain from use from 7 days prior to the first dose and throughout the study.
* Is using a proton pump inhibitor and cannot refrain from use from 7 days prior to the first dose and throughout the study.
* Is using a sensitive substrate of P-gp with a narrow therapeutic window (e.g. digoxin).
* Any other condition, including significant skin or nail disease, that in the opinion of the Investigator would place the patient at an unacceptable risk or cause the patient to be unlikely to fully participate or comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 2: Incidence of Treatment-emergent Adverse Events (TEAEs) | Up to 4.5 years
Part 1 and Part 2: Incidence of Adverse Events of Special Interest (AESIs) | Up to 4.5 years
Part 1 and Part 2: Incidence of Serious Adverse Events (SAEs) | Up to 4.5 years
Part 2: Objective Response Rate | Up to 4.5 years

SECONDARY OUTCOMES:
Part 1: Progression-free Survival (PFS) | Up to 4.5 years
Part 1: Objective Response Rate of NX-019 | Up to 4.5 years
Part 1 and Part 2: Plasma Concentration of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Cerebrospinal Fluid (CSF) Concentration of NX-019 | Up to 43 days
Part 1 and Part 2: Maximum Observed Serum Concentration (Cmax) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Area Under the Concentration Versus Time Curve (AUC) Over a Dosing interval (AUCtau) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: AUC from Time 0 to the Time of Last Quantifiable Plasma Concentration (AUC0-t) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: AUC from Time 0 to Infinity (AUC0-inf) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Percent of AUC Extrapolated (AUC%extrap) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Terminal Phase Elimination Half-life (t½) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Terminal Phase Elimination Rate Constant (λz) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Apparent Plasma Clearance (CL/F) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Apparent Volume of Distribution (Vd/F) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Accumulation Index Using Cmax (AICmax) and Accumulation Index Using AUC (AIAUC0-inf) of NX-019 | Day 1, 2, and 15 of Cycle 1, Day 1 and 15 of Cycle 2, Day 1 of Cycle 3 and every odd-numbered Cycle thereafter (1 Cycle is 28 days)
Part 1 and Part 2: Time to Response (TTR) | Up to 4.5 years
Part 1 and Part 2: Duration of Response (DOR) | Up to 4.5 years
Part 1 and Part 2: Disease Control Rate (DCR) | Up to 4.5 years
Part 1 and Part 2: Overall Survival (OS) | Up to 4.5 years
Part 1 and Part 2: Objective Response Rate for CNS (central nervous system) Metastases | Up to 4.5 years
Part 1 and Part 2: TTR for CNS (central nervous system) Metastases | Up to 4.5 years
Part 1 and Part 2: DOR for CNS (central nervous system) Metastases | Up to 4.5 years

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - City of Hope - Seacliff, Huntington Beach, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - HealthPartners Frauenshuh Cancer Center, Saint Louis Park, Minnesota
  - HealthPartners Cancer Center at Regions Hospital, Saint Paul, Minnesota
  - University Of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - NEXT Virginia, Fairfax, Virginia
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- National Taiwan University Cancer Center, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following final analysis.
Access Criteria: Nalo will review on a case by case basis.